CLINICAL TRIAL: NCT07081061
Title: A Feasibility Randomized Controlled Trial Evaluating the Effectiveness of a Digital Mental Health Intervention for Moderate/Severe Depression and Anxiety
Brief Title: Clinical Outcomes of a Digital Mental Health Intervention for Moderate/Severe Depression and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teladoc Health (Industry)
Collaborators: BetterHelp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BH2294015
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Depression, Anxiety; Mental Health Issue; Mental Health Wellness 2
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants enrolled in a digital mental health platform, which provided access to licensed therapists, group therapy sessions, and a library of educational articles.
  Interventions: Other: BetterHelp
- Control (No Intervention): Participants were not enrolled in a digital mental health platform, but continued their standard routine or care as needed.

INTERVENTIONS:
Other: BetterHelp — Use program as needed for 16 weeks
  Arms: Intervention

SUMMARY:
A digital mental health intervention (BetterHelp, Mountain View, CA) provides users with access to online therapy care for treatment of depression and anxiety. This feasibility randomized controlled trial compares clinical outcomes of an intervention group, who will enroll in the digital mental health platform, to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Has moderate or severe baseline anxiety or depression, as defined by GAD-7 ≥ 10 or PHQ-9 ≥ 10, respectively
* Based in the US
* Fluent in the English language
* Has an email account to receive and complete online surveys
* Has access to a smartphone, tablet or computer
* Able to understand and provide informed consent

Exclusion Criteria:

* Pregnant or plan on becoming pregnant in the next 6 months
* Has no or mild baseline anxiety or depression, as defined by GAD-7 < 10 and PHQ-9 < 10, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 90 days
  Recruitment rates for study participation
Adherence | 90 days
  Adherence rates to study procedures

SECONDARY OUTCOMES:
GAD-7 | Baseline, 45 days, 90 days
  Anxiety will be measured by the Generalized Anxiety Disorder Scale (GAD-7), ranging from 0 (no anxiety) to 21 (severe anxiety). The percentage of participants who achieved a minimal clinically important difference (MCID) of 4 points or more will also be reported for each group, as based on literature.
PHQ-9 | Baseline, 45 days, 90 days
  Depression will be measured by the Patient Health Questionnaire (PHQ-9), ranging from 0 (no depression) to 27 (severe depression). The percentage of participants who achieved a minimal clinically important difference (MCID) of 5 points or more will also be reported for each group, as based on literature.

OTHER OUTCOMES:
Workplace Productivity | Baseline, 45 days, 90 days
  Workplace productivity will be measured by the Work Productivity and Activity Impairment Questionnaire (WPAI) and reported for both groups.
Sleep | Baseline, 45 days, 90 days
  Sleep quality will be measured by the Jenkins Sleep Scale (JSS-4) and reported for both groups.
Stress | Baseline, 45 days, 90 days
  Stress levels will be measured by the Perceived Stress Scale (PSS-10) and reported for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Hong, PhD, Principal Investigator — Teladoc Health

IPD SHARING:
Plan to Share IPD: No